CLINICAL TRIAL: NCT07062081
Title: Correlation Between Acne Vulgaris and Lipid Profile Among Young Adults in Sohag Governorate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hager Ali Dardier, demonostrator at family medicine department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-25-06-18MS
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: lipid profile — The blood samples were taken to measure lipid profile levels as triglycerides (TG), total cholesterol (TC), low-density lipoprotein cholesterol (LDL), and high-density lipoprotein cholesterol (HDL) and VLDL values.

SUMMARY:
Acne vulgaris is the most common skin condition affecting late adolescents worldwide.1 The prevalence of acne is said to be 85% in adults aged 12 to 25 years.2 Almost all teenagers between 15 and 17 years report having some degree of acne.3 Estimates of the lifetime occurrence of acne in the literature range from 0.1%4 to as high as 85.1%5 in the general population, depending on the age range, region, and method of sampling. Overall, acne is more common in women,8,9 but in some literature the prevalence is approximately equal in men and women.10,11

DETAILED DESCRIPTION:
Acne vulgaris is a multifactorial disorder of the pilosebaceous unit, resulting from sebum overproduction, follicular hyperkeratinization, inflammation, and bacterial colonization of hair follicles by Propionibacterium acnes. The sebaceous gland is controlled primarily by hormonal stimulation. In this way, the hormonal effect on sebum secretion is a key to the pathogenesis of acne.12-16 During puberty, alteration of the sebum component, called dysseborrhea, stress, irritation, cosmetics, and potential dietary factors lead to the formation of acne lesions.16 Changes in sebum secretion are considered to be an important factor of acne. In this way, increased sebum secretion can induce acne occurrence.17 Increasing evidence, in essence, indicates that changes in lipid profile are strongly related to acne occurrence. Accordingly, further information and awareness campaigns are needed to emphasize the role of balanced lipid metabolism to control acne. Although a correlation between the incidence of acne and lipid profile levels has been observed before, it must be documented in each population with etiological characteristics. Minimal reports are available on the relationship between plasma lipids and acne in our country. Hence, we aim to establish this study to estimate the presence of lipid alteration in acne patients.

ELIGIBILITY:
Inclusion Criteria:

* age- and sex-matched healthy volunteers, not taking any medicine, and having no personal or family history of acne.

Exclusion Criteria:

* : reluctance to take part in the study, pregnancy or lactation

  * intake of oral contraception or hormone therapy, history of taking any medications that affect lipid metabolism or oral isotretinoin
  * and systemic diseases that affect the metabolism of lipids, such as uncontrolled diabetes, hypothyroidism, nephrotic syndrome, end-stage renal failure, HIV, familial hypercholesterolemia, and metabolic syndrome.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
lipid profile (TG) | 6 months
  The blood samples were taken to measure lipid profile levels as triglycerides (TG)
lipid profile (HDL) | 6 months
  The blood samples were taken to measure lipid profile levels as HDL
lipid profile (VLDL) | 6 months
  The blood samples were taken to measure lipid profile levels as VLDL

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Degitz K, Ochsendorf F. Pharmacotherapy of acne. Expert Opin Pharmacother. 2008 Apr;9(6):955-71. doi: 10.1517/14656566.9.6.955. PMID 18377339
- [Background] Gibbs S. Skin disease and socioeconomic conditions in rural Africa: Tanzania. Int J Dermatol. 1996 Sep;35(9):633-9. doi: 10.1111/j.1365-4362.1996.tb03687.x. PMID 8876289
- [Background] Dreno B. Treatment of adult female acne: a new challenge. J Eur Acad Dermatol Venereol. 2015 Jun;29 Suppl 5:14-9. doi: 10.1111/jdv.13188. PMID 26059821
- [Background] Collier CN, Harper JC, Cafardi JA, Cantrell WC, Wang W, Foster KW, Elewski BE. The prevalence of acne in adults 20 years and older. J Am Acad Dermatol. 2008 Jan;58(1):56-9. doi: 10.1016/j.jaad.2007.06.045. Epub 2007 Oct 22. PMID 17945383